CLINICAL TRIAL: NCT04831125
Title: Conduction System Pacing International Registry (CONSPIRE)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB20-1601
Record Dates: First submitted 2021-03-15; First posted 2021-04-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bradyarrhythmia; Heart Failure
Keywords: Conduction system pacing (CSP); His bundle pacing (HBP); Left ventricular septal pacing (LVS); Left bundle branch area pacing (LBBAP); Proximal left conduction system pacing (LCS)
MeSH Terms: conditions — Bradycardia; Heart Failure | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals receiving conduction system pacing
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection on the use of pacemaker, implantable cardioverter-defibrillator (ICD), and cardiac resynchronization therapy (CRT) devices and leads that are approved for clinical use.

SUMMARY:
The purpose of this registry study is to collect information about routine clinical practices with device implantation to treat bradycardia and cardiac systolic dysfunction (heart rhythm disorders) across global centers of excellence in cardiac pacing. In particular, this study will examine the use of conduction system pacing (CSP) in clinical practice. Information collected in the registry will help researchers better characterize strengths and limitations of current technology and treatments.

DETAILED DESCRIPTION:
During this past decade, there has been a dramatic surge in interest in new physiologic pacing strategies which engage and take advantage of the intrinsic cardiac conduction system. These approaches include His bundle pacing (HBP) as well as approaches which seek to pace the proximal left conduction system (LCS), including left bundle branch area pacing (LBBAP) or pacing in the region of the left posterior fascicle. Left ventricular septal pacing (LVS) has also been proposed as another means to avoid dyssynchrony with early data suggestive of comparable electrical synchronization as biventricular pacing. These approaches utilize approved pacing systems and leads which are delivered to new targets in the His-Purkinje system or LV endocardial fibers. Despite the growing interest in HBP, LCS, and LVS, the majority of data are from disparate cohort studies and there has been a lack of uniformity in assembling data or analyzing and interpreting outcomes.

The goal of the Conduction System Pacing International Registry (CONSPIRE) is to systematically and prospectively collect data across multiple centers of excellence on the early implementation of permanent conduction system pacing devices in order to characterize strengths and limitations of current technology. The study will evaluate patient selection, intraprocedural characteristics, and clinical outcomes among patients receiving conduction system pacing (CSP) as part of their routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Meets American College of Cardiology (ACC)/American Heart Association (AHA)/Heart Rhythm Society (HRS) guidelines for bradycardia, or
* Meets ACC/AHA/HRS guidelines for cardiac resynchronization therapy (CRT).

Exclusion Criteria:

* Age < 18 years
* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Pregnancy
* Difficulty with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals receiving conduction system pacing
  * Any presence of symptomatic bradyarrhythmia requiring pacing therapy
  * Any presence of heart failure (HF) with evidence of wide QRS or anticipated requirement for >40% ventricular pacing
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Implant characteristics | Month 0, during procedure
  Data will be collected on CSP lead position based on reported anatomical position (e.g., His bundle location, left bundle branch area or left bundle branch pacing location, or left ventricular septal pacing location)
QRS duration measured by electrocardiography at baseline | Baseline, within 1 month prior to procedure
  Data will be collected on QRS duration (milliseconds) prior to implant
QRS morphology captured by surface electrocardiography at baseline | Baseline, within 1 month prior to procedure
  Data will be collected on QRS morphology (e.g., narrow QRS, left bundle branch block, right bundle branch block, left anterior or posterior hemiblock, nonspecific intraventricular conduction delay, or predominantly paced QRS) prior to implant
QRS duration measured by electrocardiography after implant | Month 0, pre discharge
  Data will be collected on QRS duration (milliseconds) after implant procedure
QRS morphology captured by surface electrocardiography after implant | Month 0, pre discharge
  Data will be collected on QRS morphology [e.g., narrow QRS, left bundaloid QRS in V1, or right bundaloid QRS in V1] after implant procedure
Procedure-related complications | Through 12 months
  Data will be collected to characterize procedure-related complications
Changes in left ventricular ejection fraction | Through 12 months
  Data will be collected to characterize changes in left ventricular ejection fraction
Changes in chamber dimension | Through 12 months
  Data will be collected to characterize changes in chamber dimension
Heart failure hospitalizations | Through 12 months
  Data will be collected to characterize heart failure hospitalizations within the first 12 months after device implant
Any-cause mortalities | Through 12 months
  Data will be collected to characterize any-cause mortalities within the first 12 months after device implant
Sustained ventricular arrhythmia occurrences | Through 12 months
  Data will be collected to characterize sustained ventricular arrhythmia occurrences
System-related complications | Through 12 months
  Data will be collected to characterize system-related complications
Lead-related complications | Through 12 months
  Data will be collected to characterize lead-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav A Upadhyay, MD, Principal Investigator — University of Chicago
Locations (8):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - University of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai & Mount Sinai Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
- Maastricht University Medical Center, Maastricht, Netherlands
- Health Research Institute Hospital La Fe, Valencia, Spain
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No